CLINICAL TRIAL: NCT01999634
Title: Evaluation of Microdialysis to Monitor Postoperative Outcomes After Proctectomy
Brief Title: Monitoring by Microdialysis of Postoperative Complications After Proctectomy
Acronym: MTM-COLON-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2012_843_0024; 2013-A00261-44 (Other: ID-RCB)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer
Keywords: rectum; microdialysis; anastomotic leaks
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cma microdialysis catheter placement (Experimental): At the end of the surgery the cma microdialysis catheter is placed near the anastomosis
  Interventions: Device: cma microdialysis catheter placement

INTERVENTIONS:
Device: cma microdialysis catheter placement — the microdialysis catheters are sold by CMA

SUMMARY:
The aim of this study is to monitor by microdialysis the postoperative outcomes in order to identify anastomotic leaks after rectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* rectal disease requiring proctectomy with anastomosis and stomy
* proctectomy by laparoscopy or laparotomy
* written consent

Exclusion Criteria:

* history of colorectal surgery
* rectal surgery without anastomosis
* breastfeeding or pregnancy
* ASA score IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
anastomotic leaks rate | postoperative day 30
  the anastomotic leaks rate is defined as the number of anastomotic leaks validated by a CT scan or at the clinical examination

SECONDARY OUTCOMES:
superficial surgical site infection rate | postoperative day 30
  the surgical site infection rate is defined as the number of infection near the incision
functional success of microdialysis | postoperative day 5
  the functional success of microdialysis is defined as abnormal values localised at the microdialysis catheter

CONTACTS AND LOCATIONS:
Overall Officials: jean marc regimbeau, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- Amiens university hospital, Amiens, France

REFERENCES:
- [Background] Solligard E, Juel IS, Spigset O, Romundstad P, Gronbech JE, Aadahl P. Gut luminal lactate measured by microdialysis mirrors permeability of the intestinal mucosa after ischemia. Shock. 2008 Feb;29(2):245-51. doi: 10.1097/SHK.0b013e3180cab3ce. PMID 17693938
- [Background] Cibicek N, Zivna H, Zadak Z, Kulir J, Cermakova E, Palicka V. Colon submucosal microdialysis: a novel in vivo approach in barrier function assessment - a pilot study in rats. Physiol Res. 2007;56(5):611-617. doi: 10.33549/physiolres.931004. Epub 2006 Dec 19. PMID 17184153
- [Background] Krejci V, Hiltebrand L, Buchi C, Ali SZ, Contaldo C, Takala J, Sigurdsson GH, Jakob SM. Decreasing gut wall glucose as an early marker of impaired intestinal perfusion. Crit Care Med. 2006 Sep;34(9):2406-14. doi: 10.1097/01.CCM.0000233855.34344.29. PMID 16878039
- [Result] Beauchemin M, Gonzalez-Frankenberger B, Tremblay J, Vannasing P, Martinez-Montes E, Belin P, Beland R, Francoeur D, Carceller AM, Wallois F, Lassonde M. Mother and stranger: an electrophysiological study of voice processing in newborns. Cereb Cortex. 2011 Aug;21(8):1705-11. doi: 10.1093/cercor/bhq242. Epub 2010 Dec 13. PMID 21149849